CLINICAL TRIAL: NCT03301220
Title: A Phase 3 Randomized, Multicenter Study of Subcutaneous Daratumumab Versus Active Monitoring in Subjects With High-Risk Smoldering Multiple Myeloma
Brief Title: A Study of Subcutaneous Daratumumab Versus Active Monitoring in Participants With High-Risk Smoldering Multiple Myeloma
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR108172; 54767414SMM3001 (Other: Janssen Research & Development, LLC); 2016-001205-16 (EudraCT Number); 2023-507143-11-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2017-09-29; First posted 2017-10-04 (Actual); Results first posted 2025-12-23 (Actual); Last update posted 2026-01-30 (Actual); Status verified 2026-01

CONDITIONS: Smoldering Multiple Myeloma
MeSH Terms: conditions — Smoldering Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A: Active Monitoring (No Intervention): Participants randomized to active monitoring will receive no study medication, but will undergo the same disease evaluations at the same frequency as participants randomized to daratumumab.
- Arm B: Daratumumab SC (Experimental): Participants will receive 1800 milligram (mg) of daratumumab co-formulated with 2000 units per milliliter (U/mL) of recombinant human hyaluronidase (rHuPH20) by subcutaneous (SC) injection until 39 cycles or up to 36 months or until confirmed disease progression, unacceptable toxicity or withdrawal from the study treatment, study termination or study completion.
  Interventions: Drug: Daratumumab SC: daratumumab + rHuPH20

INTERVENTIONS:
Drug: Daratumumab SC: daratumumab + rHuPH20 — Participants will receive daratumumab SC injection (daratumumab 1800 mg + rHuPH20 [2000 U/mL]) once weekly for Cycles 1 and 2 (Days 1, 8, 15, and 22 of each week), every 2 weeks for Cycle 3 to Cycle 6 (Days 1 and 15), and thereafter every 4 weeks (Day 1) until 39 cycles or up to 36 months or until confirmed disease progression, unacceptable toxicity or withdrawal from the study treatment, study termination or study completion. Each cycle is 28 days in duration.
  Other Names: JNJ-54767414
  Arms: Arm B: Daratumumab SC

SUMMARY:
The primary objective of this study is to determine whether treatment with daratumumab administered subcutaneously (SC) prolongs progression-free survival (PFS) compared with active monitoring in participants with high-risk smoldering multiple myeloma (SMM).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of high risk smoldering multiple myeloma (SMM) (per International Myeloma Working Group [IMWG] criteria) for less than or equal to (<=) 5 years with measurable disease at the time of randomization, defined as serum M protein greater than or equal to (>=) 10 gram per liter (g/L) or urine M protein >= 200 milligram per 24 hours (mg/24 hours) or involved serum free light chain (FLC) >=100 milligram per liter (mg/L) and abnormal serum FLC ratio
* Clonal bone marrow plasma cells (BMPCs) >= 10 percentage (%); and at least 1 of the following risk factors; Serum M protein >= 30 g/L, immunoglobulin (Ig)A SMM, immunoparesis with reduction of 2 uninvolved immunoglobulin isotypes (only IgA, IgM, and IgG should be considered in determination for immunoparesis; IgD and IgE are not considered in this assessment), serum involved: uninvolved FLC ratio >= 8 and less than (<) 100, or clonal BMPCs greater than (>) 50% to <60% with measurable disease
* Eastern Cooperative Oncology Group (ECOG) performance status score of 0 or 1
* Women of childbearing potential must commit to either abstain continuously from heterosexual sexual intercourse or to use highly effective method of contraception
* A woman of childbearing potential must have a negative serum or urine pregnancy test at screening within 14 days prior to randomization
* During the study and for 3 months after receiving the last dose of daratumumab, a woman must agree not to donate eggs (ova, oocytes) for the purposes of assisted reproduction

Exclusion Criteria:

* Multiple myeloma (MM), requiring treatment, defined by any of the following:

  1. Bone lesions (1 or more osteolytic lesions on low-dose whole body computed tomography [LDCT], positron-emission tomography with computed tomography [PET-CT] or CT). Participants who have benign/post-traumatic bone lesions visible on screening images as well as previous imaging, may be considered for inclusion. Details (diagnosis, location, duration) on benign/post-traumatic pre-existing bone lesions that can be seen on the screening images (example [eg.], old fractures) and were also present on previous imaging are to be reported in the case report form (CRF)
  2. Hypercalcemia (serum calcium greater than [>]0.25 millimoles per liter [mmol/L] [>1 milligram per deciliter {mg/dL}] higher than upper limit of normal [ULN] or >2.75 mmol/L [>11 mg/dL]). Participants who have clinically stable hypercalcemia attributable to a disease other than multiple myeloma (eg, hyperparathyroidism) may be considered for inclusion after a case by case review by the medical monitor
  3. Renal insufficiency, preferably determined by creatinine clearance less than (<)40 milliliter per minute (mL/min) measured or estimated using the Modification of Diet in Renal Disease (MDRD), or serum creatinine >177 micromole per liter (μmol/L). Participants who have clinically stable renal insufficiency attributable to a disease other than multiple myeloma (eg, glomerulonephritis) may be considered for inclusion after a case by case review by the medical monitor
  4. Anemia, defined as hemoglobin <10 gram per deciliter (g/dL) or >2 g/dL below lower limit of normal or both; transfusion support or concurrent treatment with erythropoietin stimulating agents is not permitted. Participants who have clinically stable anemia attributable to a disease other than multiple myeloma (eg, thalassemia, vitamin B12 deficiency, iron deficiency) may be considered for inclusion after a case by case review by the medical monitor
  5. Clonal BMPC percentage >=60%
  6. Serum FLC ratio (involved:uninvolved) >=100 (the involved FLC must be >=100 mg/L)
  7. More than 1 focal lesion >=5 millimeter (mm) in diameter by magnetic resonance imaging (MRI)
* Primary systemic amyloid light-chain (AL) (immunoglobulin light chain) amyloidosis
* Exposure to any of the following:

  1. Prior exposure to daratumumab or prior exposure to other anti-Cluster of Differentiation 38 (anti-CD38) therapies
  2. Prior exposure to approved or investigational treatments for SMM or MM (including but not limited to conventional chemotherapies, immunomodulatory agent [IMiDs], or proteasome inhibitor [PIs]). Stable standard dosing of bisphosphonate and denosumab as indicated for osteoporosis is acceptable
  3. Exposure to investigational drug (including investigational vaccines) or invasive investigational medical device for any indication within 4 weeks or 5 half-lives, whichever is longer, before Cycle 1, Day 1
  4. Ongoing treatment with corticosteroids with a dose >10 milligram (mg) prednisone or equivalent per day at the time of randomization; or >280 mg cumulative prednisone dose or equivalent for any 4-week period in the year prior to randomization
  5. Ongoing treatment with other monoclonal antibodies (eg, infliximab, rituximab), immunomodulators (eg, abatacept, methotrexate, azathioprine, cyclosporine) or other treatments that are likely to interfere with the study procedures or results
* Received treatment (chemotherapy, surgery, et cetera [etc]) for a malignancy (other than SMM) within 3 years before the date of randomization (exceptions are squamous and basal cell carcinomas of the skin, carcinoma in situ of the cervix or breast, or other non-invasive lesion), which is considered cured with minimal risk of recurrence within 3 years
* Medical or psychiatric condition or disease (for example, active systemic disease [including presence of auto-antibodies], uncontrolled diabetes) that is likely to interfere with the study procedures or results, or that in the opinion of the investigator, would constitute a hazard for participating in this study
* Known allergies, hypersensitivity, or intolerance to corticosteroids, monoclonal antibodies, hyaluronidase, or other human proteins, or their excipients, or known sensitivity to mammalian-derived products (including dairy allergy)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 390 (Actual)
Dates: Start 2017-11-07 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2026-06-30 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (163):
- United States (23):
  - Arizona Oncology Associates, PC - HAL, Phoenix, Arizona
  - Innovative Clinical Research Inc, Whittier, California
  - Miami Cancer Institute, Miami, Florida
  - Emory University, Atlanta, Georgia
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - East Jefferson General Hospital, Metairie, Louisiana
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Mayo Clinic, Rochester, Minnesota
  - Washington University, St Louis, Missouri
  - VA Southern Nevada Healthcare, North Las Vegas, Nevada
  - New York Oncology Hematology, Albany, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - University of North Carolina, Chapel Hill, North Carolina
  - Levine Cancer Institute, Carolinas HealthCare System, Charlotte, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
  - The Ohio State University, Columbus, Ohio
  - OHSU/CHM, Portland, Oregon
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Texas Oncology P A, Austin, Texas
  - VA North Texas Health Care System, Dallas, Texas
  - Texas Oncology P A, Tyler, Texas
  - University of Washington, Seattle, Washington
- Argentina (6):
  - Hospital Aleman, Buenos Aires
  - Hospital Italiano de Buenos Aires, Buenos Aires
  - CEMIC Saavedra, Ciudad de Buenos Aires
  - Hospital Privado Centro Medico de Cordoba, Córdoba
  - Hospital Italiano de La Plata, La Plata
  - Sanatorio Britanico de Rosario, Rosario
- Australia (4):
  - Austin Hospital, Heidelberg
  - Calvary Mater Newcastle Hospital, Waratah
  - The Perth Blood Institute, West Perth
  - Queen Elizabeth Hospital, Woodville
- Belgium (6):
  - ZNA, Antwerp
  - AZ St.-Jan Brugge-Oostende AV, Bruges
  - UZBrussel, Brussels
  - UZ Gent, Ghent
  - Virga Jessa Ziekenhuis, Hasselt
  - Az Groeninge, Kortrijk
- Brazil (10):
  - Centro de Pesquisa e Ensino em Oncologia de Santa Catarina CEPEN, Florianópolis
  - Universidade Federal de Goias - Hospital das Clinicas da UFG, Goiânia
  - Instituto Joinvilense de Hematologia e Oncologia Ltda Centro de Hematologia e Oncologia, Joinville
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Instituto de Educacao, Pesquisa e Gestao em Saude Instituto Americas (COI), Rio de Janeiro
  - Hospital Sao Rafael, Salvador
  - Fundacao Faculdade Regional de Medicina de Sao Jose do Rio Preto Hospital de Base, São José do Rio Preto
  - Instituto de Ensino e Pesquisa São Lucas, São Paulo
  - Clinica Sao Germano, São Paulo
  - Hospital Santa Cruz, São Paulo
- Canada (3):
  - Arthur J E Child Comprehensive Cancer Centre, Calgary, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Lakeridge Health Oshawa, Oshawa, Ontario
- Czechia (4):
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - Fakultni Nemocnice Ostrava, Ostrava
  - Fakultni nemocnice Plzen, Hemato-onkologicke oddeleni, Pilsen
  - Vseobecna fakultni nemocnice v Praze - I. interni klinika - klinika hematologie, Prague
- Denmark (4):
  - Ålborg Universitetshospital, Aalborg
  - Aarhus University Hospital, Aarhus N
  - Rigshospitalet, Copenhagen
  - Odense Universitetshospital, Odense C
- France (7):
  - CHU de Limoges - Fédération Hépatologie, Limoges
  - Chu Hotel Dieu, Nantes
  - CHU de Bordeaux - Hospital Haut-Leveque, Pessac
  - Centre hospitalier Lyon-Sud, Pierre-Bénite
  - CHU De Poitiers, Poitiers
  - l'Hôpital Pontchaillou, Rennes
  - CHU Bretonneau, Tours
- Germany (6):
  - Helios Kliniken Berlin Buch Gmbh, Berlin
  - St. Barbara-Klinik Hamm GmbH, Hamm
  - Universitaetsklinikum Heidelberg Medizinische Klinik V, Heidelberg
  - Medizinische Klinik A, Münster
  - Universitaetsklinikum Tuebingen der Eberhard-Karls-Universitaet, Abteilung fuer Innere Medizin II,, Tübingen
  - Universitaetsklinikum Ulm, Ulm
- Alexandra General Hospital of Athens, Athens Attica, Greece
- Hungary (4):
  - Semmelweis Egyetem, I. Belgyogyaszati Klinika, Budapest
  - Semmelweis Egyetem I.Belgyogyaszati Klinika, Budapest
  - Del Pesti Centrumkorhaz Orszagos Hematologiai es Infektologiai Intezet Szent Laszlo Telephely, Budapest
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- Israel (10):
  - Haemek, Afula
  - Barzilai Medical Center, Ashkelon
  - Bnai Zion Medical Center, Haifa
  - Carmel Medical Center, Haifa
  - Rambam Medical Center, Haifa
  - Hadassah Medical Center, Jerusalem
  - Galilee Medical Center, Nahariya
  - Rabin Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Sourasky Medical Center, Tel Aviv
- Italy (7):
  - Policlinico Sant'Orsola Malpighi, Bologna
  - Businco Cancer Hospital, Cagliari
  - A.O. Santa Croce e Carle, Cuneo
  - Ospedale S. Eugenio, Roma
  - Università di Roma 'La Sapienza' - Ospedale Umberto 1°, Roma
  - A.O.U. Città della Salute e della Scienza di Torino- Divisione di Ematologia, Torino
  - ASST dei Sette Laghi, Ospedale di Circolo e Fonazione Macchi, Varese
- Japan (18):
  - Fukuoka University Hospital, Fukuoka
  - Chugoku Central Hospital, Fukuyama
  - Ogaki Municipal Hospital, Gifu
  - Kagoshima University Hospital, Kagoshima
  - Kanazawa University Hospital, Kanazawa
  - National Hospital Organization Osaka Minami Medical Center, Kawachi-Nagano
  - Kobe City Medical Center General Hospital, Kobe
  - National Hospital Organization Kumamoto Medical Center, Kumamoto
  - Kurume University Hospital, Kurume
  - Kyoto Kuramaguchi Medical Center, Kyoto
  - National Hospital Organization Matsumoto Medical Center, Matsumoto
  - Matsuyama Red Cross Hospital, Matsuyama
  - Nagoya City University Hospital, Nagoya
  - Niigata Cancer Center Hospital, Niigata
  - National Hospital Organization Okayama Medical Center, Okayama
  - National Hospital Organization Sendai Medical Center, Sendai
  - National Hospital Organization Shibukawa Medical Center, Shibukawa
  - Japanese Red Cross Medical Center, Shibuya City
- Mexico (5):
  - iBiomed Research Unit, Aguascalientes
  - JM Research, SC, Cuernavaca
  - Centro de Investigación Farmacéutica Especializada, Guadalajara
  - Centro de Atención e Investigación Clínica en Oncología, Mérida
  - Hospital Universitario de Nuevo León, Monterrey
- Netherlands (4):
  - Gelre Ziekenhuis, Apeldoorn
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - Haga ziekenhuis, The Hague
  - ETZ TweeSteden, Tilburg
- Oslo University Hospital HF Ulleval sykehus, Oslo, Norway
- Poland (5):
  - Szpital Specjalistyczny w Brzozowie Podkarpacki Osrodek Onkologiczny im Ks B Markiewicza, Brzozów
  - Szpital Uniwersytecki nr 2 im. Jana Biziela w Bydgoszczy, Bydgoszcz
  - Wojewodzki Szpital Specjalistyczny w Legnicy, Legnica
  - Clinical Research Center Sp z o o Medic R Sp k, Poznan
  - Instytut Hematologii i Transfuzjologii, Warsaw
- Russia (9):
  - Emergency Hospital of Dzerzhinsk, Dzerzhinsk
  - City clinical hospital n.a. S.P.Botkin, Moscow
  - City Clinical Hospital # 40, Moscow
  - Nizhniy Novgorod Region Clinical Hospital, Nizhny Novgorod
  - Perm Medical Sanitary Unit#1, Perm
  - Republican Hospital n.a.V.A.Baranov, Petrozavodsk
  - Ryazan Regional Clinical Hospital, Ryazan
  - Clinical Research Institute of Hematology and Transfusiology, Saint Petersburg
  - Oncology Dispensary of Komi Republic, Syktyvkar
- Spain (10):
  - Hosp. Univ. Germans Trias I Pujol, Badalona
  - Hosp Clinic de Barcelona, Barcelona
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Gral. Univ. Gregorio Maranon, Madrid
  - Hosp. Univ. Infanta Leonor, Madrid
  - Hosp. Univ. Ramon Y Cajal, Madrid
  - Clinica Univ. de Navarra, Pamplona
  - Hosp. Quiron Madrid Pozuelo, Pozuelo de Alarcón
  - Hosp Clinico Univ de Salamanca, Salamanca
  - Hosp. Univ. Dr. Peset, Valencia
- Sweden (3):
  - Falu Lasarett, Falun
  - Sunderby Sjukhus Medicinkliniken, Luelå
  - Karolinska Universitetssjukhuset Huddinge, Stockholm
- Turkey (Türkiye) (6):
  - Ankara Numune Egitim ve Arastirma Hastanesi, Ankara
  - Ankara University Medical Faculty, Ankara
  - Trakya University Hospital, Edirne
  - Istanbul University Istanbul Medical Faculty, Istanbul
  - Erciyes University Medical Faculty, Kayseri
  - Ondokuz Mayis University, Samsun
- United Kingdom (7):
  - Heart of England NHS Foundation Trust, Birmingham
  - University Hospitals Bristol NHS Trust, Bristol
  - Kent and Canterbury Hospital, Canterbury
  - St Bartholomew's Hospital, London
  - Christie Hospital NHS Trust, Manchester
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Royal Stoke University Hospital, Stoke-on-Trent

REFERENCES:
- [Derived] Dimopoulos MA, Voorhees PM, Schjesvold F, Cohen YC, Hungria V, Sandhu I, Lindsay J, Baker RI, Suzuki K, Kosugi H, Levin MD, Beksac M, Stockerl-Goldstein K, Oriol A, Mikala G, Garate G, Theunissen K, Spicka I, Mylin AK, Bringhen S, Uttervall K, Pula B, Medvedova E, Cowan AJ, Moreau P, Mateos MV, Goldschmidt H, Ahmadi T, Sha L, Cortoos A, Katz EG, Rousseau E, Li L, Dennis RM, Carson R, Rajkumar SV; AQUILA Investigators. Daratumumab or Active Monitoring for High-Risk Smoldering Multiple Myeloma. N Engl J Med. 2025 May 8;392(18):1777-1788. doi: 10.1056/NEJMoa2409029. Epub 2024 Dec 9. PMID 39652675

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Results are currently reported until the primary completion date (01 May 2024). Results of remaining duration will be posted upon study completion.
Groups:
- Arm A: Active Monitoring (ACTM): Participants in the active monitoring group did not receive any study medication but underwent disease evaluations for every 12 weeks until disease progression (PD) as those randomized to receive daratumumab.
- Arm B: Daratumumab SC: Participants received daratumumab 1800 milligrams (mg) co-formulated with recombinant human hyaluronidase (rHuPH20) 2000 units per milliliter (U/mL) as subcutaneous (SC) injection once every week (Q1W) (Days 1, 8, 15, and 22 of each week) in Cycles 1 and 2, every 2 weeks (Q2W) (Days 1 and 15) from Cycle 3 to Cycle 6, and thereafter every 4 weeks (Day 1) from Cycle 7 to Cycle 39, for a maximum of 36 months, or until confirmed disease progression, unacceptable toxicity or withdrawal from the study treatment. In addition, disease evaluations were performed every 12 weeks until PD. Each treatment cycle was 28 days. After end of treatment, participants were followed up for safety until death, lost to follow up, consent withdrawal or study end, whichever occurred first (up to 8 years).
Period: Overall Study
Arm/Group | Arm A: Active Monitoring (ACTM) | Arm B: Daratumumab SC
Started | 196 | 194
Treated | 196 | 193
Completed | 0 | 0
Not Completed | 196 | 194
Not completed — Death | 26 | 15
Not completed — Withdrawal by Subject | 23 | 12
Not completed — Lost to Follow-up | 1 | 1
Not completed — Randomized in error | 1 | 1
Not completed — Randomized but not treated | 0 | 1
Not completed — Ongoing followup | 145 | 163
Not completed — Principal Investigator and participant decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Active Monitoring (ACTM) | Arm B: Daratumumab SC | Total
Number analyzed (Participants) | 196 | 194 | 390
Age, Continuous [Mean (Standard Deviation); unit: Years] | 63.0 (10.76) | 61.9 (11.17) | 62.4 (10.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 99 | 202
  Male | 93 | 95 | 188
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 9 | 14 | 23
  Not Hispanic or Latino | 176 | 169 | 345
  Unknown or Not Reported | 11 | 11 | 22
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 3 | 0 | 3
  Asian | 13 | 18 | 31
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 2
  Black or African American | 7 | 4 | 11
  White | 162 | 161 | 323
  More than one race | 0 | 1 | 1
  Unknown or Not Reported | 9 | 10 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  Belgium | 6 | 4 | 10
  France | 9 | 7 | 16
  Germany | 4 | 4 | 8
  Netherlands | 6 | 3 | 9
  United States | 27 | 30 | 57
  Argentina | 5 | 4 | 9
  Australia | 10 | 5 | 15
  Brazil | 3 | 8 | 11
  Canada | 6 | 2 | 8
  Czech Republic | 2 | 6 | 8
  Denmark | 0 | 2 | 2
  Greece | 3 | 8 | 11
  Hungary | 8 | 4 | 12
  Israel | 28 | 28 | 56
  Italy | 4 | 8 | 12
  Japan | 13 | 15 | 28
  Norway | 8 | 7 | 15
  Poland | 6 | 6 | 12
  Russian Federation | 9 | 4 | 13
  Spain | 14 | 10 | 24
  Sweden | 3 | 2 | 5
  Turkey | 5 | 9 | 14
  United Kingdom | 17 | 18 | 35

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS) as Assessed by the Independent Review Committee (IRC)
Description: PFS was defined as the duration from the date of randomization to either progressive to multiple myeloma (MM), according to the International Myeloma Working Group (IMWG) diagnostic criteria for MM, or death due to any cause, whichever occurred first. Per IMWG criteria, active MM by SLiM-CRAB defined as: greater than or equal to (>=) 60 percent (%) bone marrow plasma cells (BMPCs), free light chain (FLC) involved/uninvolved ratio >=100, greater than (>)1 focal bone lesions on magnetic resonance imaging (MRI), calcium elevation, renal insufficiency by creatinine clearance, anemia, or bone disease due to lytic bone lesions. Kaplan-Meier estimate was used.
Time Frame: From randomization (Day -5) up to 77 months
Population: Intent-to-treat (ITT) analysis set included all participants randomized into the study.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Arm A: Active Monitoring (ACTM) | Arm B: Daratumumab SC
Number analyzed (Participants) | 196 | 194
Months | 41.46 [26.41 to 53.32] | NA [66.69 to NA] — Here "NA" signifies that median and upper limit of 95% confidence interval (CI) were not estimable due to low number of participants with events.
Statistical Analysis 1: Comparison: Arm A: Active Monitoring (ACTM) vs Arm B: Daratumumab SC; Test type: Superiority; p < 0.0001, Log Rank; Hazard Ratio (HR) = 0.49, 95% CI 2-sided [0.36 to 0.67]

2. Secondary Outcome: Time to Biochemical or Diagnostic (SLiM-CRAB) Progression Per Computerized Algorithm Analyses
Time Frame: From randomization (Day -5) up to 8 years
Reporting Status: Not Posted, anticipated posting 2027-01

3. Secondary Outcome: Overall Response Rate (ORR)
Time Frame: From randomization (Day -5) up to 8 years
Reporting Status: Not Posted, anticipated posting 2027-01

4. Secondary Outcome: Complete Response (CR) Rate
Time Frame: From randomization (Day -5) up to 8 years
Reporting Status: Not Posted, anticipated posting 2027-01

5. Secondary Outcome: Time to First-Line Treatment for Multiple Myeloma
Time Frame: From randomization (Day -5) up to 8 years
Reporting Status: Not Posted, anticipated posting 2027-01

6. Secondary Outcome: Progression-Free Survival on First-Line Treatment for Multiple Myeloma (PFS2)
Time Frame: From randomization (Day -5) up to 8 years
Reporting Status: Not Posted, anticipated posting 2027-01

7. Secondary Outcome: Best Response on First-line Therapy for Multiple Myeloma
Time Frame: From randomization (Day -5) up to 8 years
Reporting Status: Not Posted, anticipated posting 2027-01

8. Secondary Outcome: Overall Survival (OS)
Time Frame: From randomization (Day -5) up to 8 years
Reporting Status: Not Posted, anticipated posting 2027-01

9. Secondary Outcome: Percentage of Participants Who Progressed to Multiple Myeloma With Adverse Prognostic Features
Time Frame: From randomization (Day -5) up to 8 years
Reporting Status: Not Posted, anticipated posting 2027-01

10. Secondary Outcome: Maximum Observed Serum Concentration (Cmax) of Daratumumab
Time Frame: Cycles 1 and 3 : Day 1 predose, and Day 4 postdose; Cycles 5, 7, 12, and 24: Day 1 predose; end of the treatment (EOT, 37.11 months); and 8 weeks after the last daratumumab dose (up to 38.11 months). Each Cycle was 28 days
Reporting Status: Not Posted, anticipated posting 2027-01

11. Secondary Outcome: Minimum Observed Serum Concentration (Cmin) of Daratumumab
Time Frame: Cycles 1 and 3 : Day 1 predose, and Day 4 postdose; Cycles 5, 7, 12, and 24: Day 1 predose; EOT( 37.11 months); and 8 weeks after the last daratumumab dose (up to 38.11 months). Each Cycle was 28 days
Reporting Status: Not Posted, anticipated posting 2027-01

12. Secondary Outcome: Number of Participants With Anti-daratumumab Antibodies
Time Frame: Cycles 1 and 3 : Day 1 predose, and Day 4 postdose; Cycles 5, 7, 12, and 24: Day 1 predose; EOT (37.11 months); and 8 weeks after the last daratumumab dose (up to 38.11 months). Each Cycle was 28 days
Reporting Status: Not Posted, anticipated posting 2027-01

13. Secondary Outcome: Number of Participants With Anti-Recombinant Human Hyaluronidase (rHuPH20) Antibodies
Time Frame: Cycles 1, 3, 5, 7, 12, and 24 : Predose on Day 1; EOT (37.11 months); and 8 weeks after the last daratumumab dose (up to 38.11 months). Each Cycle was 28 days
Reporting Status: Not Posted, anticipated posting 2027-01

14. Secondary Outcome: Change From Baseline in European Organization for Research and Treatment of Cancer Quality of Life Questionnaire (EORTC QLQ-C30) Score
Time Frame: From Baseline (Day -35) up to 8 years
Reporting Status: Not Posted, anticipated posting 2027-01

15. Secondary Outcome: Change From Baseline in the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire for Patients With Multiple Myeloma (EORTC QLQ-MY20) Future Perspective Scale
Time Frame: From Baseline (Day -35) up to 8 years
Reporting Status: Not Posted, anticipated posting 2027-01

16. Secondary Outcome: Change From Baseline in European Quality (EuroQoL) 5-Dimension 5-Level Health Status (EQ-5D-5L) Questionnaire Score
Time Frame: From Baseline (Day -35) up to 8 years
Reporting Status: Not Posted, anticipated posting 2027-01

17. Secondary Outcome: Duration of Response
Time Frame: From randomization (Day -5) up to 8 years
Reporting Status: Not Posted, anticipated posting 2027-01

18. Secondary Outcome: Time to Response
Time Frame: From randomization (Day -5) up to 8 years
Reporting Status: Not Posted, anticipated posting 2027-01

ADVERSE EVENTS:
Time Frame: All-cause mortality: From randomization (Day -5) up to 77 months, Serious adverse events (SAE) and other adverse events (AEs): active monitoring Arm : From start of treatment (Cycle 1 Day 1) up to 37 months; daratumumab SC arm: From start of treatment (Cycle 1 Day 1) up to 30 days after the last dose of study treatment (up to 37.11 months)
Description: All Cause Mortality: all participants randomized into the study; SAEs and Other AEs: Safety analysis set included all randomized participants for participants randomized to active monitoring or all randomized participants who received at least one dose of daratumumab for participants randomized to daratumumab.
Arm/Group | Arm A: Active Monitoring (ACTM) | Arm B: Daratumumab SC
All-Cause Mortality (participants affected / at risk) | 26/196 | 15/194
Serious Adverse Events (participants affected / at risk) | 38/196 | 56/193
Other Adverse Events (participants affected / at risk) | 140/196 | 178/193
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Active Monitoring (ACTM) (N=196) | Arm B: Daratumumab SC (N=193)
Iron Deficiency Anaemia (Blood and lymphatic system disorders) | 1 | 1
Angina Pectoris (Cardiac disorders) | 1 | 1
Atrial Fibrillation (Cardiac disorders) | 0 | 1
Cardiac Arrest (Cardiac disorders) | 1 | 0
Cardiac Failure (Cardiac disorders) | 1 | 0
Myocardial Ischaemia (Cardiac disorders) | 2 | 0
Sinus Tachycardia (Cardiac disorders) | 0 | 1
Hypoacusis (Ear and labyrinth disorders) | 1 | 0
Vertigo Positional (Ear and labyrinth disorders) | 0 | 1
Cataract (Eye disorders) | 0 | 1
Glaucoma (Eye disorders) | 1 | 0
Lacrimation Increased (Eye disorders) | 0 | 1
Abdominal Pain (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 2
Dysphagia (Gastrointestinal disorders) | 0 | 1
Haemorrhoidal Haemorrhage (Gastrointestinal disorders) | 1 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1
Inguinal Hernia (Gastrointestinal disorders) | 0 | 2
Intestinal Obstruction (Gastrointestinal disorders) | 0 | 1
Obstruction Gastric (Gastrointestinal disorders) | 1 | 0
Small Intestinal Obstruction (Gastrointestinal disorders) | 1 | 2
Volvulus (Gastrointestinal disorders) | 0 | 1
Chest Pain (General disorders) | 1 | 0
Gait Disturbance (General disorders) | 0 | 1
Non-Cardiac Chest Pain (General disorders) | 0 | 2
Pain (General disorders) | 1 | 0
Pelvic Mass (General disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 1
Cholecystitis (Hepatobiliary disorders) | 2 | 0
Cholecystitis Acute (Hepatobiliary disorders) | 0 | 1
Appendicitis (Infections and infestations) | 1 | 0
Bacteraemia (Infections and infestations) | 1 | 0
Cellulitis (Infections and infestations) | 0 | 2
Corneal Infection (Infections and infestations) | 0 | 1
Covid-19 (Infections and infestations) | 0 | 3
Covid-19 Pneumonia (Infections and infestations) | 1 | 2
Diverticulitis (Infections and infestations) | 1 | 1
Erysipelas (Infections and infestations) | 0 | 1
Gastroenteritis Norovirus (Infections and infestations) | 0 | 1
Lower Respiratory Tract Infection (Infections and infestations) | 0 | 1
Metapneumovirus Infection (Infections and infestations) | 0 | 1
Pharyngitis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 1 | 7
Pneumonia Bacterial (Infections and infestations) | 1 | 1
Pneumonia Pneumococcal (Infections and infestations) | 1 | 0
Pneumonia Streptococcal (Infections and infestations) | 0 | 1
Pneumonia Viral (Infections and infestations) | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 2
Sepsis (Infections and infestations) | 2 | 2
Septic Arthritis Staphylococcal (Infections and infestations) | 0 | 1
Septic Shock (Infections and infestations) | 1 | 1
Sinusitis (Infections and infestations) | 0 | 1
Urinary Tract Infection (Infections and infestations) | 1 | 1
Vestibular Neuronitis (Infections and infestations) | 1 | 0
West Nile Viral Infection (Infections and infestations) | 0 | 1
Ankle Fracture (Injury, poisoning and procedural complications) | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1
Femoral Neck Fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip Fracture (Injury, poisoning and procedural complications) | 0 | 1
Humerus Fracture (Injury, poisoning and procedural complications) | 0 | 1
Incisional Hernia (Injury, poisoning and procedural complications) | 0 | 1
Rib Fracture (Injury, poisoning and procedural complications) | 1 | 2
Shoulder Fracture (Injury, poisoning and procedural complications) | 0 | 1
Spinal Compression Fracture (Injury, poisoning and procedural complications) | 2 | 1
Splenic Injury (Injury, poisoning and procedural complications) | 1 | 0
Subdural Haematoma (Injury, poisoning and procedural complications) | 0 | 1
Traumatic Fracture (Injury, poisoning and procedural complications) | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Intervertebral Disc Protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Breast Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Invasive Ductal Breast Carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Neoplasm of Appendix (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Plasmacytoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Brain Oedema (Nervous system disorders) | 0 | 1
Cerebellar Stroke (Nervous system disorders) | 1 | 0
Cerebral Ischaemia (Nervous system disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 0
Intracranial Aneurysm (Nervous system disorders) | 0 | 1
Ischaemic Stroke (Nervous system disorders) | 1 | 0
Transient Ischaemic Attack (Nervous system disorders) | 0 | 1
Abortion Spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 | 0
Acute Kidney Injury (Renal and urinary disorders) | 2 | 0
Haematuria (Renal and urinary disorders) | 1 | 0
Renal Injury (Renal and urinary disorders) | 1 | 0
Benign Prostatic Hyperplasia (Reproductive system and breast disorders) | 1 | 0
Pelvic Organ Prolapse (Reproductive system and breast disorders) | 1 | 0
Acute Respiratory Failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Chronic Obstructive Pulmonary Disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Emphysema (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Organising Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pulmonary Embolism (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary Oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dermal Cyst (Skin and subcutaneous tissue disorders) | 0 | 1
Diabetic Foot (Skin and subcutaneous tissue disorders) | 0 | 1
Neurodermatitis (Skin and subcutaneous tissue disorders) | 0 | 1
Breast Prosthesis Removal (Surgical and medical procedures) | 0 | 1
Radical Prostatectomy (Surgical and medical procedures) | 0 | 1
Deep Vein Thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm A: Active Monitoring (ACTM) (N=196) | Arm B: Daratumumab SC (N=193)
Anaemia (Blood and lymphatic system disorders) | 19 | 9
Neutropenia (Blood and lymphatic system disorders) | 5 | 13
Palpitations (Cardiac disorders) | 1 | 13
Cataract (Eye disorders) | 6 | 10
Abdominal Pain (Gastrointestinal disorders) | 12 | 18
Abdominal Pain Upper (Gastrointestinal disorders) | 0 | 12
Constipation (Gastrointestinal disorders) | 8 | 18
Diarrhoea (Gastrointestinal disorders) | 9 | 51
Dyspepsia (Gastrointestinal disorders) | 2 | 10
Gastrooesophageal Reflux Disease (Gastrointestinal disorders) | 2 | 12
Nausea (Gastrointestinal disorders) | 9 | 37
Vomiting (Gastrointestinal disorders) | 7 | 16
Asthenia (General disorders) | 15 | 18
Chest Discomfort (General disorders) | 2 | 10
Fatigue (General disorders) | 26 | 66
Influenza Like Illness (General disorders) | 7 | 17
Injection Site Erythema (General disorders) | 0 | 31
Oedema Peripheral (General disorders) | 3 | 20
Pyrexia (General disorders) | 4 | 33
Bronchitis (Infections and infestations) | 5 | 13
Covid-19 (Infections and infestations) | 10 | 15
Influenza (Infections and infestations) | 1 | 10
Nasopharyngitis (Infections and infestations) | 23 | 49
Pneumonia (Infections and infestations) | 9 | 17
Sinusitis (Infections and infestations) | 5 | 17
Upper Respiratory Tract Infection (Infections and infestations) | 15 | 58
Urinary Tract Infection (Infections and infestations) | 10 | 12
Contusion (Injury, poisoning and procedural complications) | 3 | 10
Fall (Injury, poisoning and procedural complications) | 12 | 10
Arthralgia (Musculoskeletal and connective tissue disorders) | 35 | 52
Back Pain (Musculoskeletal and connective tissue disorders) | 38 | 46
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 1 | 12
Myalgia (Musculoskeletal and connective tissue disorders) | 9 | 20
Pain in Extremity (Musculoskeletal and connective tissue disorders) | 15 | 28
Dizziness (Nervous system disorders) | 8 | 19
Headache (Nervous system disorders) | 13 | 35
Paraesthesia (Nervous system disorders) | 8 | 17
Peripheral Sensory Neuropathy (Nervous system disorders) | 3 | 16
Anxiety (Psychiatric disorders) | 7 | 14
Insomnia (Psychiatric disorders) | 5 | 43
Cough (Respiratory, thoracic and mediastinal disorders) | 12 | 33
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 10 | 29
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 3 | 18
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 3 | 16
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 2 | 11
Alopecia (Skin and subcutaneous tissue disorders) | 1 | 10
Erythema (Skin and subcutaneous tissue disorders) | 0 | 17
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 17
Rash (Skin and subcutaneous tissue disorders) | 1 | 16
Flushing (Vascular disorders) | 0 | 10
Hypertension (Vascular disorders) | 19 | 20

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the Sponsor for review at least 60 days before submission for publication or presentation. If requested by the Sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2024-09-23): https://cdn.clinicaltrials.gov/large-docs/20/NCT03301220/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-16): https://cdn.clinicaltrials.gov/large-docs/20/NCT03301220/SAP_001.pdf